CLINICAL TRIAL: NCT06981767
Title: Effect of Topical Bromelain Versus Topical Corticosteroids in the Management of Oral Lichen Planus : A Randomized Clinical Trial
Brief Title: Effect of Topical Bromelain Versus Topical Corticosteroids in the Management of Oral Lichen Planus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lujain Taleb Suleiman Aladwan, Master's Student in Oral Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 325
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Bromelains; Triamcinolone Acetonide; Orabase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical Bromelain in Orabase (Experimental): Participants in this group will receive topical bromelain incorporated into an orabase.
  Patients will be instructed to apply the formulation four times daily No additional topical medications will be permitted.
  Interventions: Dietary Supplement: Topical Bromelain
- Topical Triamcinolone Acetonide in Orabase (Active Comparator): This group will receive topical 0.1% triamcinolone acetonide The treatment will be applied four times daily, following the same instructions and precautions as in Arm 1
  Interventions: Drug: 0.1% topical triamcinolone acetonide
- Combination of Topical Bromelain and Triamcinolone Acetonide in Orabase (Experimental): Participants in this arm will be treated with a combination formulation containing both topical bromelain and 0.1% triamcinolone acetonide in orabase.
  Application instructions will be identical to those in the other arms: four times daily.
  Interventions: Combination Product: Combination of Topical Bromelain and Triamcinolone Acetonide in Orabase

INTERVENTIONS:
Dietary Supplement: Topical Bromelain — A natural enzyme-based formulation derived from pineapple, bromelain in orabase is being investigated for its anti-inflammatory and wound-healing properties. As a non-steroidal alternative, it offers a potentially safer treatment option with minimal side effects.
  Arms: Topical Bromelain in Orabase
Drug: 0.1% topical triamcinolone acetonide — A corticosteroid-based standard treatment for OLP, triamcinolone acetonide in orabase is used for its strong anti-inflammatory and immunosuppressive effects. It serves as the conventional treatment versus novel therapy in this study
  Arms: Topical Triamcinolone Acetonide in Orabase
Combination Product: Combination of Topical Bromelain and Triamcinolone Acetonide in Orabase — This novel formulation combines the enzymatic, healing properties of bromelain with the anti-inflammatory property of triamcinolone. It is designed to provide enhanced therapeutic effects through synergistic action, potentially reducing the required corticosteroid dose while improving clinical outcomes.
  Arms: Combination of Topical Bromelain and Triamcinolone Acetonide in Orabase

SUMMARY:
Bromelain, an enzyme extract derived from pineapples, has shown promise due to its anti-inflammatory and wound-healing properties. However, its efficacy in treating oral mucosal ulcers remains unexplored. This study aims to provide clinical evidence on the efficacy of bromelain for managing OLP, potentially offering a safer and more effective treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from symptomatic OLP
* Patients free from any visible oral lesions other than OLP.
* Patients who agreed to take the supplied interventions.
* Patient who will agree to participate in the study.
* Patients who will accept to sign the informed consent.

Exclusion Criteria:

* Patients suffering from any systemic disease.
* Treatment with any systemic treatment such as systemic steroids, other immunosuppressive drugs or non-steroidal anti-inflammatory drugs at least eight weeks.
* Treatment with any oral topical medications for at least four weeks prior to the study.
* Pregnant and lactating mothers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | Recorded at baseline, and weekly for 4 weeks
  Clinical improvement will be measured using Thongprasom et al. scoring system. In Thongprasom et al. scale, lesions are given score as follows: 0, no lesions, normal mucosa; 1, Mild white striae, no erythematous area; 2, White striae with atrophic area < 1 cm2; 3, White striae with atrophic area > 1 cm2; 4, White striae with erosive area < 1 cm2 and 5, White striae with erosive area > 1 cm2 (Thongprasom et al., 2003).

SECONDARY OUTCOMES:
Pain intensity | baseline, daily for the first week, then weekly for the remaining 3 weeks.
  Pain intensity will be measured using Visual analogue scale (VAS), VAS is a self-reported pain score ranging from 0 to 10 (Cheng et al., 2012) at baseline, daily for the first week, then weekly for the remaining 3 weeks.
Oral health-related quality of life | at baseline, and weekly for the 4 weeks.
  Oral health-related quality of life using Oral Health Impact Profile-14 (OHIP-14) Oral health-related quality of life is a five-point Likert-type scale used in scoring each item of the OHIP-14. Responses are coded 0 = never', 1 = hardly ever', 2 = occasionally', 3 = fairly often', 4 = very often'. Item responses are summed to produce an OHIP-14 total score. Total OHIP-14 scores range from 0 (no impact) to 56 (all of the oral health problems are experienced very often). High scores indicates a poor oral health-related quality of life (Wiriyakijja et al., 2018).